CLINICAL TRIAL: NCT01284127
Title: Phase IV Observational Study of Deferiprone (Ferriprox®) in the Treatment of Superficial Siderosis
Brief Title: Observational Study of Deferiprone (Ferriprox®) in the Treatment of Superficial Siderosis
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00067749
Record Dates: First submitted 2011-01-20; First posted 2011-01-26 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Superficial Siderosis
Keywords: superficial siderosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deferiprone: All patients must have MRI evidence of superficial siderosis and be treated with deferiprone according to standard of care guidelines.

SUMMARY:
Superficial siderosis is a progressive neurological disease caused by iron deposition in the central nervous system (CNS) from chronic subarachnoid bleeding. Until 2011, there has been no effective treatment for this progressive condition that leads to hearing loss, spasticity, weakness, loss of bowel/bladder function, incoordination, dementia and ultimately death.

Last year, the investigators demonstrated that a lipid soluble iron chelator, deferiprone, can reduce hemosiderin deposition in patients with superficial siderosis by MRI in as little as 3 months. As the only therapy that can improve this condition, chelation with deferiprone is the standard of care for treatment of superficial siderosis. Now that the FDA has approved deferiprone in the United States for thalassemia, the investigators propose documenting the clinical effect of deferiprone over 2 years in superficial siderosis patients. The investigators' goal is to understand how the clinical course of this disease is altered using standard of care chelation therapy with deferiprone.

Patients with superficial siderosis who are taking deferiprone for chelation therapy at doses consistent with the standard of care will be offered enrollment into this observational study. Patients will be treated and monitored locally by participating neurologists who have agreed to help the investigators collect information for this study. The investigators are interested in documenting the clinical effect of deferiprone on hearing, ataxia and myelopathy using standardized scales performed and documenting the effect of deferiprone on hemosiderin deposition in the CNS by MRI, all performed according to standard of care.

DETAILED DESCRIPTION:
First described over 100 years ago, superficial siderosis is a rare neurodegenerative disease caused by iron toxicity in the CNS due to chronic subarachnoid bleeding. Iron from red blood cells in the subarachnoid space is preferentially taken up by the Bergmann glia in the cerebellum, brainstem, spinal cord, eighth cranial nerve and the cerebral cortex; the iron is stored as ferritin within the glial cells. With continued subarachnoid bleeding, the glia are overwhelmed by the ferritin load and die. Glial cell loss exposes neurons to free iron which is toxic to cells because it catalyzes the breakdown of hydrogen peroxide to superoxide, a reactive oxygen species that can cause lipid peroxidation, membrane dysfunction, and neuronal cell death.

Neurological consequences of iron overload depend on the area of the brain exposed to free iron. With chronic subarachnoid bleeding, the blood tends to pool around the brainstem, cerebellum and spinal cord thus leading to the classic triad of hearing loss, ataxia and myelopathy that is seen in more than 50% of patients with superficial siderosis. The eighth cranial nerve courses through the subarachnoid space until it reaches the inner ear exposing it to the toxic blood; in contrast, the other cranial nerves are protected by the peripheral Schwann cells within 1 mm of exiting the brainstem. Compared to the other CNS structures affected in superficial siderosis, the eighth cranial nerve is the most susceptible because it exposes the most surface area to volume. Thus, the most common and often the first symptom patients get is sensorineural hearing loss. This is followed by ataxia due to dysfunction of both the vestibular component of the eighth cranial nerve and neurodegeneration of the cerebellum. Myelopathy develops when the brainstem and spinal cord are involved. With continued bleeding, other areas of the brain can degenerate leading to a myriad of other symptoms seen in superficial siderosis including urinary problems headaches, anosmia, diplopia, bowel problems, ageusia, cranial nerve palsies, and dementia.

The etiologies of chronic subarachnoid bleeding are (in order of incidence): Idiopathic, Head/back trauma, A/V malformations, Current CNS tumor, Previously resected CNS tumor, CNS post-surgical (non-tumor), Amyloid angiopathy, Brachial plexus/root injury. Currently, there are fewer than 50 patients world-wide with the diagnosis of superficial siderosis. In the United States, there are an estimated 50-60 patients.

Iron chelators, other than deferiprone, used in other iron-overload disorders such as hemochromatosis are not expected to be effective in superficial siderosis because iron chelators do not cross the blood brain barrier. Copper chelators used in Wilson's disease can permeate the brain-blood barrier, but are unfortunately not effective in superficial siderosis, as copper chelators do not bind iron. Surgical intervention is thought to be key to slowing the disease by stanching the leak of blood into the subarachnoid space. However, once the neurodegenerative process has begun, surgical intervention does not prevent the neurodegenerative disease from progressing.

Recently, the investigators have demonstrated that deferiprone, a lipid-soluble iron chelator, at a dose of 30 mg/kg/day administered over 90 days is safe in a population of 10 superficial siderosis patients. Although not designed to assess efficacy, the investigators also found that 4 of 10 patients showed reduced hemosiderin deposition in the CNS after the trial, which is very different from the natural course of disease in which hemosiderin deposition either remains the same over 3 months or increases over time. This suggests that deferiprone may be effective in chelating hemosiderin in patients with superficial siderosis.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of superficial siderosis by MRI.
2. Must be receiving deferiprone according to standard of care under the supervision of the treating physician.
3. Must be able to understand and sign the informed consent form.

Exclusion Criteria:

1. If the patient is unwilling or unable to comply with the requirements of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with MRI-confirmed superficial siderosis currently residing in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2018-01-08 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levy M, Llinas RH. Deferiprone reduces hemosiderin deposits in the brain of a patient with superficial siderosis. AJNR Am J Neuroradiol. 2011 Jan;32(1):E1-2. doi: 10.3174/ajnr.A2331. Epub 2010 Nov 4. PMID 21051507

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deferiprone
Started | 38
Completed | 31
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Deferiprone
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38
Cause of Bleed [Count of Participants; unit: Participants]
  Dural Tear | 11
  Prior Neurosurgical Procedure | 8
  Central Nervous System (CNS) Tumor/Cyst | 4
  Undetermined | 15
Duration of Clinical Disease [Median (Full Range); unit: years] | 7 [1 to 33]
Participants with Repair of Bleed [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Show Stability, Improvement or Decline in Self Reported Hearing
Description: Number of participants who show stability, improvement or decline in self reported hearing.
Time Frame: At the end of the 2-year period
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone
Number analyzed (Participants) | 31
Participants
  Stable | 13
  Worse | 18
  Improved | 0

2. Primary Outcome: Number of Participants Who Show Stability, Improvement or Decline in Self Reported Coordination
Description: Number of participants who show stability, improvement or decline in self reported coordination.
Time Frame: At the end of the 2-year period
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone
Number analyzed (Participants) | 31
Participants
  Stable | 8
  Worse | 21
  Improved | 2

3. Primary Outcome: Number of Participants Who Show Stability, Improvement or Decline in Self Reported Walking
Description: Number of participants who show stability, improvement or decline in self reported walking.
Time Frame: At the end of the 2-year period
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone
Number analyzed (Participants) | 31
Participants
  Stable | 9
  Worse | 21
  Improved | 1

4. Primary Outcome: Number of Participants Who Show Stability, Improvement or Decline in Self Reported Fine Motor Function
Description: Number of participants who show stability, improvement or decline in self reported fine motor function.
Time Frame: At the end of the 2-year period
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone
Number analyzed (Participants) | 31
Participants
  Stable | 9
  Worse | 22
  Improved | 0

5. Primary Outcome: Number of Participants Who Show Stability, Improvement or Decline in Self Reported Bowel/Bladder Function
Description: Number of participants who show stability, improvement or decline in self reported bowel/bladder function.
Time Frame: At the end of the 2-year period
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone
Number analyzed (Participants) | 31
Participants
  Stable | 12
  Worse | 18
  Improved | 1

6. Secondary Outcome: Number of Participants With MRI of the Brain and Spinal Cord Showing Changes in Hemosiderin Deposition
Description: MRI of the brain and spinal cord without contrast to monitor for changes in hemosiderin deposition in terms of worsening or improvement.
Time Frame: Baseline, At the end of the 2-year period
Population: All participants with follow up MRIs (16) were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone
Number analyzed (Participants) | 16
Participants
  Worse | 8
  Improved | 8

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Deferiprone
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 10/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferiprone (N=38)
Fatigue (Nervous system disorders) | 10 — Self reported fatigue
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 — Self reported joint pain
Mouth sores (Skin and subcutaneous tissue disorders) | 2 — Self reported mouth sores

LIMITATIONS AND CAVEATS:
The major limitations of this study relate to the observational design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT01284127/Prot_SAP_000.pdf